CLINICAL TRIAL: NCT07372599
Title: Influence of Therapeutic Failure on the Psychosocial Experience of Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Influence of Therapeutic Failure on the Psychosocial Experience in Multiple Sclerosis
Acronym: INPSYSEP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Lille (Other); Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL) - France (Unknown); Centre Hospitalier Universitaire, Amiens (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A01541-48
Record Dates: First submitted 2025-12-16; First posted 2026-01-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Patient-reported-outcome; Patient-reported-experience; Quality of life; Socioeconomic status; Therapeutic failure; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Occurrence of Therapeutic Failure: Occurrence of Therapeutic Failure : Change or discontinuation of the DMT decided by the treating neurologist, linked to a progression of the disease characterised by inflammatory activity (clinical and/or radiological) and/or progression of the disease unrelated to inflammatory activity.
  Interventions: Other: Questionnaires
- Absence of Therapeutic Failure
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — At inclusion (T0), TE if event occurs and T1: Completion of 5 questionnaires (MusiQoL, HADS, ICECAP-A, iPCQ, MusiCare).

SUMMARY:
Multiple sclerosis (MS), an inflammatory, neurodegenerative disease of the central nervous system, affects around 120,000 patients in France and is the leading cause of non-traumatic disability in young adults. It affects patients' health-related quality of life (QoL) and has a significant economic impact on patients and society as a whole. Early initiation of disease-modifying therapy (DMT) is recommended in relapsing-remitting MS (RRMS). Nevertheless, according to a recent French cohort, 30% of patients initially treated with a first-line FT will switch to a highly effective compound within 5 years due to its ineffectiveness. Therapeutic failure (Th-F) is therefore a frequent occurrence, but its psychological, social and economic consequences are poorly understood. These elements are generally the subject of measurements reported by patients, and several studies have highlighted the importance of taking them into account in the management of these patients.

Here, the investigators will study two categories of these measures in a Th-F situation. On the one hand, patient-reported outcome measurements (PROMs) will be examined. Patients' psychological distress and their QoL are two important examples of psychosocial impacts in patients with MS, compared to the general population. The impact on activity levels is also well known, but the specific effect of Th-F has not yet been studied. On the other hand, patients' experiences of their care pathway and their opinion on the quality of care (patient-reported experience measurement [PREM]) will also be studied. Some PREMs refer to care coordination, satisfaction with the relationship with carers or doctors' empathy levels. To date, data on the experience of MS patients regarding their care pathway remains limited and non-existent during Th-F.

Finally, the influence of socioeconomic status (SES) on PROMs and PREMs is worth considering. In the general population, patients' experience of care can be influenced by their socioeconomic status. Compared with research on other diseases (notably cardiovascular diseases and cancers), there is relatively little work on the association between socioeconomic status and MS and none has focused on the topic of Th-F.

The investigators therefore hypothesise that a quality of care perceived favourably by MS patients may moderate the negative impact of Th-F on their QoL, anxiety/depression and activity levels (as recently described in oncology), and a more recent measure of abilities assessing well-being defined in a broad sense, as a function of their SES.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over.
* Patient with RRMS according to McDonald 2024 criteria.
* Uninterrupted use of a moderately effective treatment, or highly effective treatment only if it is the first DMT, for at least 6 months.
* Collection of non-objection.
* Patient affiliated to the social security system.

Exclusion Criteria:

* Patient with progressive MS.
* Patient treated continuously with the same DMT for 3 years or more.
* Patient who received a second line DMT or an immunosuppressant before taking a first line DMT.
* Patients who have received mitoxantrone as the first treatment
* Pregnant or breast-feeding woman at the time of inclusion.
* Severe cognitive and/or psychological disorders which, according to the investigator (with or without a neuropsychological assessment), prevent the participant from completing the self-questionnaires independently and accurately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RRMS patients aged 18 or over with uninterrupted use of a moderately effective treatment, or highly effective treatment only if it is the first DMT, for at least 6 months.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life : The International Multiple Sclerosis Quality of Life Questionnaire (MusiQoL) | 2 years
  The International Multiple Sclerosis Quality of Life Questionnaire (MusiQoL) is a multidimensional, self-administered questionnaire that has been developed internationally (including a French version). It comprises 31 questions describing nine dimensions (daily activities, psychological well-being, relationships with friends, symptoms, relationships with family, relationships with the healthcare system, emotional and sexual life, adaptation, and rejection). Each item is scored from 1 to 5. The score of each dimension is obtained by computing the mean of the item scores of the dimension. All dimension scores are linearly transformed to a 0-100 scale. A higher score indicates a higher level of health-related quality of life.

SECONDARY OUTCOMES:
Psychological distress : The Hospital Anxiety and Depression Scale (HADS) | 2 years
  The Hospital Anxiety and Depression Scale (HADS) is validated in French. It contains 14 items divided into two dimensions (anxiety and depression). Each item is scored from 0 to 3. The score for each subscale is the sum of the 7 items (ranging from 0-21). A higher score indicates a higher distress. This questionnaire has already been used with MS patients and has shown good psychometric indicators.
Well-being : The ICEpop CAPability measure for Adults (ICECAP-A) | 2 years
  The ICEpop CAPability measure for Adults (ICECAP-A) is a measure of the capability of the general adult population (18+) intended for use in economic evaluation and focused on well-being in the broad sense, rather than health. ICECAP-A comprises five attributes (attachment, stability, fulfilment, pleasure, autonomy). Each item is scored from 1 to 4. The total score is the sum of the 5 attributes (ranging 5-20). A higher score indicates a higher quality of life/capability. Qualitative and quantitative studies on the validity of ICECAP-A have been carried out and a French translation of ICECAP-A has been developed for the general population.
Activity levels: The self-administered iMTA Productivity Cost Questionnaire (iPCQ) | 2 years
  The self-administered iMTA Productivity Cost Questionnaire (iPCQ) measure the impact of the disease on market and household activities. This recently validated questionnaire, available in French, comprises 18 items, of which 9 are general questions to collect demographic information, such as age, sex and respondents' work status. iPCQ includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work.
Quality of care: MusiCare | 2 years
  MusiCare is the only French-language questionnaire specific to MS for assessing the quality of care as perceived by MS patients and their careers. It comprises 35-item encompassing 5 domains: information about the disease (11), information about the treatments/medical investigations (8), relationships with healthcare teams (8), healthcare access (5) and reception conditions in care centers (3). Each item is scored from 1 to 5. All dimension scores are linearly transformed and standardized using a scale ranging from 0 to 100. A higher score indicates a higher self-perceived care management quality.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT07372599/Prot_SAP_000.pdf